CLINICAL TRIAL: NCT02208505
Title: Antitussive Effect of Single-dose Dexmedetomidine With Low-dose Remifentanil Infusion During Emergence in Adults After Thyroidectomy: Comparison With High-dose Remifentanil Infusion Alone
Brief Title: Antitussive Effect of Single-dose Dexmedetomidine With Low-dose Remifentanil Infusion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Jeong Soo Lee, Clinical Assistant Professor, Yonsei University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 3-2013-0192'
Record Dates: First submitted 2014-02-11; First posted 2014-08-05 (Estimated); Last update posted 2017-10-18 (Actual); Status verified 2017-10

CONDITIONS: Thyroidectomy
MeSH Terms: interventions — Dexmedetomidine; Remifentanil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Dexmedetomidine (Experimental): we administrate the single-dose dexmedetomidine (0.5mcg/kg) with low-dose remifentanil infusion(TCI 1 ng/ml).
  Interventions: Drug: Dexmedetomidine + Remifentanil-low dose
- Remifentanil (Active Comparator): we administrate the high-dose remifentanil infusion(TCI 2 ng/ml) alone.
  Interventions: Drug: Remifentanil-high dose

INTERVENTIONS:
Drug: Dexmedetomidine + Remifentanil-low dose — single dose administration (0.5mcg/kg) 10 min before end of the surgery with maintain the infusion of remifentanil (TCI 1 ng/ml) until end of surgery
  Other Names: Precedex
  Arms: Dexmedetomidine
Drug: Remifentanil-high dose — maintain the infusion of remifentanil until end of the surgery (TCI 2 ng/ml)
  Other Names: Ultiva
  Arms: Remifentanil

SUMMARY:
After thyroid surgery, the incidence and severity of coughing is important because it may cause serious complications, such as bleeding in the surgical field, laryngospasm, and cardiovascular disturbance. Several studies have shown that the single-dose of dexmedetomidine is effective for reducing cough and agitation during emergence from general anesthesia.

To test the hypothesis that single-dose of dexmedetomidine combined with a low-dose remifentanil infusion during emergence from general anaesthesia could reduce coughing as good as high-dose remifentanil infusion, we will evaluate the efficacy on cough suppression and reduction of side effect of remifentanil using non-inferiority trial.

ELIGIBILITY:
Inclusion Criteria:

* Thyroid disease undergoing thyroidectomy
* age 20-65
* Amerian society of anesthesgiologist class 1 or 2

Exclusion Criteria:

* chronic cough
* difficult intubation
* liver disease
* uncontrolled hypertension

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2014-02; Primary Completion 2015-07 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Incidence of coughing during emergence from general anesthesia | from 5min before extubation to 5min after extubation

SECONDARY OUTCOMES:
side effect of remifentanil | up to 1 day after surgery
  comparison of the incidence of delayed awakening, post-operative nausea/vomiting, consumption of pain killer

OTHER OUTCOMES:
quality of recovery from anesthesia | upto 1day after surgery
  using Quality of Recovery-40 questionnaire, evaluate the recovery status of patient from general anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Soo Lee, Principal Investigator — Yonsei University
Locations (1):
- Gangnam severance hospital, Seoul, South Korea